CLINICAL TRIAL: NCT03328494
Title: A Phase 1/1b Study of Paclitaxel in Combination With BOS172722, a Monopolar Spindle 1 Kinase Inhibitor, in Patients With Advanced Nonhaematologic Malignancies
Brief Title: Study of Paclitaxel in Combination With BOS172722 in Patients With Advanced Nonhaematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boston Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BOS172722-01; 2017-001749-29 (EudraCT Number)
Record Dates: First submitted 2017-10-30; First posted 2017-11-01 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Advanced Nonhaematologic Malignancies
Keywords: Paclitaxel; BOS172722; triple-negative breast cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — BOS172722; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part A: Monotherapy (BOS172722) (Experimental): BOS172722 will be administered on Days 1, 2, 8, 9, 15, and 16 of each 28-day cycles in participants with histopathologically confirmed advanced nonhaematologic malignancies.
  Interventions: Drug: BOS172722
- Part A: Combination therapy (BOS172722 + Paclitaxel) (Experimental): BOS172722 will be administered on Cycle 0 Day 1 and on Days 1, 2, 8, 9, 15, and 16 in Cycle 1 and subsequent 28-day cycles in participants with histopathologically confirmed advanced nonhaematologic malignancies. The participants will also receive 80 milligrams per meters squared (mg/m^2) paclitaxel as an intravenous (IV) infusion on Days 1, 8, and 15 of each 28-day cycle. During dose escalation, further exploration of the treatment schedule for the BOS172722-paclitaxel combination will be initiated. In such combination cohorts, BOS172722 will be administered with paclitaxel on Days 1, 8, and 15 only of each treatment cycle (except for Cycle 2 Day1), and will not be administered on Day 2, 9, and 16. These alternative schedules will be explored to further characterize the pharmacokinetics and tolerability of such a dosing regimen.
  Interventions: Drug: BOS172722; Drug: Paclitaxel
- Part B: Combination therapy (BOS172722 + Paclitaxel) (Experimental): Participants with triple-negative breast cancer will be treated with oral BOS172722 at the recommended Phase 2 dose (RP2D) established in Part A on Days 1, 2, 8, 9, 15, and 16 of each 28-day cycle and IV paclitaxel at 80 mg/m^2 on Days 1, 8, and 15 of each 28-day cycle.
  Interventions: Drug: BOS172722; Drug: Paclitaxel

INTERVENTIONS:
Drug: BOS172722 — Oral capsules
Drug: Paclitaxel — IV infusion
  Arms: Part A: Combination therapy (BOS172722 + Paclitaxel); Part B: Combination therapy (BOS172722 + Paclitaxel)

SUMMARY:
This study will be conducted to assess the safety and tolerability of BOS172722 when administered as monotherapy and in combination with paclitaxel in participants with advanced nonhaematologic malignancies and also to establish the maximum tolerated dose and recommended Phase 2 dose of BOS172722 in combination with paclitaxel in those participants.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

* For Part A only, histopathologically confirmed diagnosis of an advanced nonhaematologic malignancy
* For Part B only, histopathologically confirmed diagnosis of triple-negative breast cancer
* No standard curative treatment or has declined standard therapy
* Eastern Cooperative Oncology Group performance status 0 or 1, measured within 72 hours before the first BOS172722 or paclitaxel dose
* Predicted life expectancy of ≥ 3 months
* Adequate renal function (creatinine ≤ 1.5 × upper limit of normal [ULN] or glomerular filtration rate ≥ 50 milliliters per minute [mL/min])
* Adequate hepatic function:

  * Total bilirubin ≤ 1.5 × ULN
  * Aspartate transaminase ≤ 3 × ULN (or ≤ 5 × ULN if due to liver involvement by tumor)
  * Alanine transaminase ≤ 3 × ULN (or ≤ 5 × ULN if due to liver involvement by tumor)
* Adequate bone marrow function:

  * Hemoglobin ≥ 9.0 grams per deciliter (g/dL)
  * Platelet count ≥ 100 × 10^9 cells per liter (cells/L)
  * Absolute neutrophil count ≥ 1.5 × 10^9 cells/L
* Mean corrected QT interval as calculated by the Fridericia correction formula < 470 milliseconds
* Willingness to use adequate contraceptive methods
* Capable of giving signed informed consent
* Willingness to avoid direct sunlight and the use of tanning equipment during the study and for at least 30 days after the last BOS172722 dose

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* For Part A combination cohorts and Part B: a history of hypersensitivity to paclitaxel
* Persistent clinically significant toxicity from prior chemotherapy > Grade 1, excluding alopecia
* Unable to swallow oral capsules
* Gastrointestinal (GI) condition which could interfere significantly with the absorption of study medication
* History of upper GI bleeding, ulceration, or perforation within 6 months before the first or paclitaxel BOS172722 dose
* Uncontrolled or severe concurrent medical condition (including uncontrolled brain metastases). (Stable brain metastases either treated or being treated with a stable dose of steroids/anticonvulsants, with no dose change within 28 days before the first BOS172722 or paclitaxel dose, will be allowed.)
* History of stroke or cerebrovascular accident within 3 months before the first BOS172722 or paclitaxel dose
* Any evidence of serious active infection
* Uncontrolled or severe cardiovascular disease, including myocardial infarct or unstable angina within 6 months before the first BOS172722 or paclitaxel dose, New York Heart Association Class II or greater congestive heart failure, serious arrhythmias requiring medication for treatment, clinically significant pericardial disease, or cardiac amyloidosis
* Uncontrolled intercurrent illness or psychiatric illness/social situations that would limit compliance with study requirements
* Known infection with Human Immunodeficiency Virus or hepatitis A, B, or C (testing not required)
* Major surgery within 28 days before the first BOS172722 or paclitaxel dose
* Pregnant or breastfeeding
* Active treatment for a secondary malignancy
* Cancer-directed therapy (chemo-, radio-, immuno-, biologic, or hormonal therapy with the exception of luteinizing hormone-releasing hormone agonists/antagonists, receptor activator of nuclear factor kappa-B ligand inhibitors, and bisphosphonates) within 21 days or 5 half-lives, whichever is longer, before the first BOS172722 or paclitaxel dose (Palliative radiotherapy is allowed before initiating study treatment if any associated toxicity resolved to ≤ Grade 1.)
* Use of a medication known to be a strong or moderate inhibitor or inducer of CYP3A4 within 14 days before the first BOS172722 or paclitaxel dose
* Use of a medication known to be a substrate of CYP3A4 and to have a narrow therapeutic range within 14 days before the first BOS172722 or paclitaxel dose
* Consumption of grapefruit or Seville oranges (including juice, marmalade, etc.) within 14 days before the first BOS172722 or paclitaxel dose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-10-13 (Actual); Primary Completion 2021-03-16 (Actual); Study Completion 2021-03-16 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | a minimum of approximately 3 months
  An AE is any untoward medical occurrence and does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of an investigational product (IP), whether or not related to the IP. AEs include pre-existing conditions that worsen.
Number of participants with a dose-limiting toxicity (DLT) | Cycle 1 (28 days)
  A DLT is defined as any toxicity attributable to BOS172722 that occurs before the end of Cycle 1.

SECONDARY OUTCOMES:
Part A Monotherapy: Plasma concentration of BOS172722 measured over 24 hours when administered alone | Cycle 1: Day 1
  The plasma concentration of BOS172722 when administered as monotherapy will be characterized
Part A Combination: Plasma concentration of BOS172722 and paclitaxel measured over 24 hours when administered either individually or in combination | Cycle 0: Day 1; Cycle 1: Day 1; Cycle 2: Day 1
  The plasma concentration of BOS172722 and paclitaxel will be characterized.
Part B Expansion: Plasma concentration of BOS172722 and paclitaxel measured over 24 hours when administered in combination | Cycle 1: Days 1 and 8 or 15
  The plasma concentration of BOS172722 and paclitaxel will be characterized.
Objective response rate (ORR) | a minimum of approximately 3 months
  ORR is defined as the percentage of participants achieving the best overall response of confirmed partial response (PR) or complete response (CR), as determined by investigator review. Responses are assessed by the Investigators using Response Evaluation Criteria in Solid Tumours (RECIST) guideline version 1.1.
Duration of response (DOR) | a minimum of approximately 3 months
  DOR is defined as the time from documentation of tumor response to disease progression. Responses are assessed by the Investigators using RECIST guideline version 1.1.
Time to response (TTR) | a minimum of approximately 3 months
  TTR is defined as the time from the start of treatment to the first objective tumor response observed for participants who achieved a CR or PR. Responses are assessed by the Investigators using RECIST guideline version 1.1.
Time to progression on study | a minimum of approximately 3 months
  Time to progression is defined as the time from treatment until objective tumor progression. This does not include deaths. Responses are assessed by the Investigators using RECIST guideline version 1.1.

CONTACTS AND LOCATIONS:
Locations (3):
- United Kingdom (3):
  - Addenbrooks Hospital, Cambridge
  - Edinburgh Cancer Centre - Western General Hospital, Edinburgh
  - Royal Marsden, London